CLINICAL TRIAL: NCT07029230
Title: Biomarker in Congenital Cardiac Surgery - sST2 Marker in Heart Failure in Congenital Heart Disease After Surgery Research and Translational Study
Brief Title: Blood Based Assessment of sST2, Taken During and After Surgery, for Pediatric Patients With Heart Defects to Predict Heart Failure.
Status: Recruiting | Type: Observational
Sponsor: Martin Schweiger (Other)
Collaborators: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor-Investigator, Martin Schweiger, Attending Physician Congenital Cardiac Surgery, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: BASEC 2024-01297; FZK 2025-INV-007 (Other: University Children's Hospital Zurich - CRC)
Record Dates: First submitted 2025-05-21; First posted 2025-06-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Congenital Heart Surgery; Congenital Heart Disease in Children; Fontan Physiology
Keywords: biomarker; sst2; congenital heart surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients planned for congenital cardiac surgery: Patients planned for congenital cardiac surgery

SUMMARY:
Patients younger than 18 scheduled for congenital heart surgery will be assessed during and post-operatively as well as at the first follow-up after 9-12 month for the novel biomarker sST2. We will assess the marker independently and in evaluation with other blood biomarkers to evaluate sings of heart failure. Compared to established biomarkers, sST2 promises thereby to be less variable to factors like age or acute kidney injury, rendering it potentially more reliable in the field of congenital cardiac surgery.

DETAILED DESCRIPTION:
Single-center prospective biomarker validation study for Soluble suppression of tumorigenicity 2 (sST2). All data will be collected upfront to ensure accuracy. The study's findings aim to improve risk stratification and guide better management for pediatric cardiac surgery patients.

Congenital Heart Disease (CHD) is the most common congenital abnormality, affecting about 1 in 100 live births. While surgical interventions have significantly improved survival rates, a considerable number of patients experience long-term complications like ventricular dysfunction and heart failure, which are major causes of death.

Biomarkers are crucial tools that can aid clinicians in risk stratification, treatment guidance, and predicting outcomes. sST2 has shown utility in adult heart surgery cases and is included in the guidelines of the American Heart Association (AHA), while it's use in pediatric cases is largely unexplored.

This study tests if sST2 as biomarker can be a useful prognostic tool for children with CHD undergoing cardiac surgery. The primary objective is to assess if a specific cut-off level of post-surgery sST2 can predict future heart failure. Secondary objectives include comparing sST2 to other established biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Consented for cardiopulmonary bypass surgery for cardiac reason
* Conversational skills in German (by child and/or representative) to be able to fully understand and sign a written consent in German language

Exclusion Criteria:

* Know genetic life limiting conditions
* Syndrome patients who are scheduled or highly likely to be operated on more than one organ
* Body weight at time of surgery less than 2.5 kg
* Being recruited and enrolled for an interventional study protocol

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients in defined age scheduled for congenital cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Surrogates of Heart Failure | 1 year post surgery
  Correlation of sST2 Levels with compound outcome of number of events of combined events of Death, need for MCS (Mechanical Circulatory Support) or Heart Transplantation

SECONDARY OUTCOMES:
30 day Mortality | 30 days after index operation
  Number of early deaths (30 days post surgery)
Overall Length of Stay | 30 days after index operation
  Time between operation and discharge from hospital
Length of intubation | 30 days after index operation
  Days necessary to wean patient from mechanical ventilatory support post surgery.
Length of Stay on ICU | 30 days after index operation
  Time between operation and discharge from the intensive care unit (ICU)
Unplanned hospital re-admission | 30 days after index operation
  Binary outcome, if patients is re-admitted for a reason related to his surgical intervention to hospital after being discharged.
Signs of upcoming heart failure, determined by cardiac echo | 30 days after index operation
  Echocardiographic signs of imminent heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schweiger, Prof, MD, MBA, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurirch, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker DM, Everett AD, Stabler ME, Jacobs ML, Jacobs JP, Vricella L, Thiessen-Philbrook H, Parikh CR, Manlhiot C, Brown JR. ST2 Predicts Risk of Unplanned Readmission Within 1 Year After Pediatric Congenital Heart Surgery. Ann Thorac Surg. 2020 Dec;110(6):2070-2075. doi: 10.1016/j.athoracsur.2020.02.056. Epub 2020 Apr 1. PMID 32246937
- [Background] Aimo A, Januzzi JL Jr, Bayes-Genis A, Vergaro G, Sciarrone P, Passino C, Emdin M. Clinical and Prognostic Significance of sST2 in Heart Failure: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Oct 29;74(17):2193-2203. doi: 10.1016/j.jacc.2019.08.1039. PMID 31648713
- [Background] Dudek M, Kaluzna-Oleksy M, Migaj J, Sawczak F, Krysztofiak H, Lesiak M, Straburzynska-Migaj E. sST2 and Heart Failure-Clinical Utility and Prognosis. J Clin Med. 2023 Apr 26;12(9):3136. doi: 10.3390/jcm12093136. PMID 37176577
- [Background] Brown JR, Stabler ME, Parker DM, Vricella L, Pasquali S, Leyenaar JK, Bohm AR, MacKenzie T, Parikh C, Jacobs ML, Jacobs JP, Everett AD. Biomarkers improve prediction of 30-day unplanned readmission or mortality after paediatric congenital heart surgery. Cardiol Young. 2019 Aug;29(8):1051-1056. doi: 10.1017/S1047951119001471. Epub 2019 Jul 10. PMID 31290383
- [Background] Maisel AS, Di Somma S. Do we need another heart failure biomarker: focus on soluble suppression of tumorigenicity 2 (sST2). Eur Heart J. 2017 Aug 7;38(30):2325-2333. doi: 10.1093/eurheartj/ehw462. No abstract available. PMID 28028009